CLINICAL TRIAL: NCT02285738
Title: Anti-Platelet and Statin Therapy to Prevent Cancer-Associated Thrombosis: A Pilot Study
Brief Title: Anti-Platelet and Statin Therapy to Prevent Cancer-Associated Thrombosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8Y14
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor; Cancer
Keywords: solid tumor, cancer, simvastatin, aspirin, blood clot, VTE, venous thromboembolism
MeSH Terms: conditions — Neoplasms; Thrombosis; Venous Thromboembolism | interventions — Aspirin; Simvastatin; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Aspirin+Asprin/Simvastatin+Observation (ASO) (Active Comparator): Aspirin 81mg/day for 4 weeks followed by 2-week washout, followed by 4 weeks of Aspirin 81mg/day with daily dose of Simvastatin with a 2-week washout period, ending with 4 weeks of observation
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation
- Aspirin+Observation+Asprin/Simvastatin (AOS) (Experimental): Aspirin 81mg/day for 4 weeks followed by 2-week washout, followed by 4 weeks of observation with 2-week washout, ending with Aspirin 81mg/day with daily dose of Simvastatin
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation
- Aspirin/Simvastatin+Observation+Asprin (SOA) (Experimental): Aspirin 81mg/day for 4 weeks with daily dose of Simvastatin followed by 2-week washout, followed by 4 weeks of observation with 2-week washout, ending with Aspirin 81mg/day
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation
- Aspirin/Simvastatin+Asprin+Observation (SAO) (Experimental): Aspirin 81mg/day for 4 weeks with daily dose of Simvastatin followed by 2-week washout, followed by 4 weeks of Aspirin 81mg/day and a 2-week washout, ending with observation for 4 weeks.
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation
- Observation+Aspirin/Simvastatin+Asprin (OSA) (Experimental): Observation for 4 weeks with 2-week washout, followed by Aspirin 81mg/day for 4 weeks with daily dose of Simvastatin followed by 2-week washout, ending with Aspirin 81mg/day for 4 weeks.
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation
- Observation+Aspirin+Asprin/Simvastatin (OAS) (Experimental): Observation for 4 weeks with 2-week washout, followed by Aspirin 81mg/day for 4 weeks followed by 2-week washout, ending with Aspirin 81mg/day for 4 weeks with daily dose of Simvastatin.
  Interventions: Drug: Aspirin; Drug: Simvastatin; Other: Observation

INTERVENTIONS:
Drug: Aspirin — 81mg/day for 4 weeks
Drug: Simvastatin — Daily dose of Simvastatin for 4 weeks
Other: Observation — participants will be observed for thrombotic evens for 4 weeks

SUMMARY:
This research study examines the safety and feasibility of aspirin with or without Simvastatin in solid tumor patients at risk for VTE (Venous Thromboembolism - or blood clots - in the arms, lets, lungs, or other part of the body). One-fifth of all thrombotic (clotting) events occur in patients that have cancer. Changes in sP-selectin will be used as a measure of efficacy. We have chosen sP-selectin as the primary marker because of its role in hemostasis, because it is predictive of thrombosis in cancer patients and because of promising preliminary data. We expect that sP-selectin levels will be elevated in patients before therapy with aspirin and/or statin, but that these levels will fall significantly during treatment, rise during the observation phase, and fall during the second study period. Patients who take part in the study have been diagnosed with a solid tumor cancer and are considered to be intermediate to high risk for VTE. The standard of care is to give chemotherapy for solid tumors and treat clots which develop using blood thinners.

DETAILED DESCRIPTION:
Objectives

Primary: To determine efficacy of aspirin with and without simvastatin in solid tumor patients at high- or intermediate-risk for VTE, in reducing markers of platelet activation, levels of inflammatory and angiogenic cytokines measured using high-throughput approaches, and clinical and investigational measures of hemostatic activation.

Secondary: To determine safety and feasibility of aspirin with or without simvastatin in solid tumor patients at high- or intermediate-risk for VTE

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignancy of a solid organ or lymphoma
* Planned to initiate a new systemic chemotherapy regimen (including patients starting on first chemotherapy or patients previously treated but starting on a new regimen)
* VTE Risk Score ≥1
* Written, informed consent.

Exclusion Criteria:

* Hematologic malignancies including acute and chronic leukemias, myelodysplastic syndromes, lymphoma and myeloma
* Primary brain tumors
* Active bleeding or high risk of bleeding in the opinion of the investigator
* Hepatic dysfunction (elevated transaminases or bilirubin > 3 times normal)
* Planned stem cell transplant
* Life expectancy < 6 months
* Acute or chronic renal insufficiency with creatinine clearance < 30 mL/min
* Pregnancy
* Known allergy to or prior intolerance of aspirin and/or simvastatin.
* Ongoing anticoagulant, statin and/or anti-platelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in average sP-selectin levels | at 16 weeks of treatment
  Change in sP-selectin levels as indicator of measure efficacy

SECONDARY OUTCOMES:
Frequency of major bleeding complications or clinically significant non-bleeding complications per patient | at 17 weeks after beginning treatment
  The safety endpoint will be bleeding complications over 17 weeks (16 weeks of study plus an additional week of observation). This will include major bleeding events and clinically significant non-major bleeding events. A bleeding event will be defined as major if it satisfies one or more of the following: decrease in hemoglobin of 2 g/dL or more, leads to transfusion of two or more units of blood or packed cells, occurs in a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial) or leads to death. Clinically significant, non-major bleeding will be defined as bleeding that does not meet the criteria for major bleeding, and has at least one of the following characteristics: multiple-source bleeding; spontaneous hematoma >25 cm2; epistaxis >5 min; macroscopic hematuria not related to instrumentation; spontaneous rectal bleeding; gingival bleeding > 5 min; hemoptysis; hematemesis; or prolonged bleeding (> 5 min) after venipuncture.
Change in average Platelet Factor 4 | at 16 weeks of treatment
  measure of efficacy using plasma level of platelet activation markers
Change in average CD40 ligand | at 16 weeks of treatment
  measure of efficacy using plasma level of platelet activation markers
Change in average serum thromboxane B2 | at 16 weeks of treatment
  measure of efficacy using plasma level of platelet activation markers
Change in average serum VEGF | at 16 weeks of treatment
  measure of efficacy using plasma level of angiogenesis markers
Change in average serum angiopoietin-2 | at 16 weeks of treatment
  measure of efficacy using plasma level of angiogenesis markers
Change in average serum hepatocyte growth factor | at 16 weeks of treatment
  measure of efficacy using plasma level of angiogenesis markers
Change in average serum PECAM | at 16 weeks of treatment
  measure of efficacy using plasma level of angiogenesis markers
Change in average serum PDGF | at 16 weeks of treatment
  measure of efficacy using plasma level of angiogenesis markers
Change in average plasma F1.2 | at 16 weeks of treatment
  measure of efficacy using plasma level of hemostatic activation markers
Change in average plasma TAT complexes | at 16 weeks of treatment
  measure of efficacy using plasma level of hemostatic activation markers
Change in average plasma D-dimer | at 16 weeks of treatment
  measure of efficacy using plasma level of hemostatic activation markers
Change in the number of thrombotic events | 17 weeks after beginning treatment
  the number of thrombotic events measured by the number of events related to venus thrombosis, pulmonary embolism, visceral vein thrombosis as well as arterial thromboembolic events including stroke, myocardial infarction or arterial embolism

CONTACTS AND LOCATIONS:
Overall Officials: Alok A Khorana, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States